CLINICAL TRIAL: NCT03245060
Title: Adapted Solution Focused Brief Therapy in Post-stroke Aphasia (SOFIA Trial): a Feasibility Study
Brief Title: Adapted Solution Focused Therapy for People With Aphasia (SOFIA Trial)
Acronym: SOFIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Staff/17-18/04; TSA Postdoc 2016/01 (Other Grant/Funding Number: The Stroke Association)
Record Dates: First submitted 2017-08-04; First posted 2017-08-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2019-01

CONDITIONS: Aphasia; Stroke
Keywords: psychosocial well-being; solution focused brief therapy
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Intervention Model Description: Wait-list control feasibility study with nested qualitative research.
  Participants will be randomly assigned to the intervention group or wait-list control group. Both groups will be assessed on psychosocial outcome measures at T1 (baseline, prior to randomisation), T2 (three months post randomisation) and T3 (six months post randomisation). Participants will also take part in in-depth interviews at T3 exploring their experiences of taking part in the project as well as complete a resource use questionnaire. All participants will receive all usual care, and up to six SFBT sessions spaced over three months delivered by Speech and Language Therapists (SLTs). The intervention group will receive the therapy immediately post randomisation, while the wait-list control group will be offered the intervention after T3. The wait-list control will additionally be reassessed at T4 (nine months post randomisation).
Who Masked: Outcomes Assessor
Masking Description: The Research Assistant will complete the psychosocial outcome measures at all time points in face to face interview format. The Research Assistant will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: immediate SFBT (Experimental): The Intervention arm will receive up to six Adapted Solution Focused Brief Therapy (SFBT) sessions immediately post randomisation. The sessions will be spaced over 3 months. Participants will also receive all usual care.
  Interventions: Behavioral: Adapted Solution Focused Brief Therapy
- Intervention: delayed SFBT (Other): The wait-list control arm will receive the same intervention (Adapted Solution Focused Brief Therapy, SFBT) as the intervention arm, but after a delay of six months. Participants will also receive all usual care.
  Interventions: Behavioral: Adapted Solution Focused Brief Therapy

INTERVENTIONS:
Behavioral: Adapted Solution Focused Brief Therapy — Solution Focused Brief Therapy is an approach to building positive change in a person's life. It builds up a picture of a client's preferred future (or how a person would like their life to be); encourages a person to notice positive signs of change; and explores personal resources, skills and resilience. In the present project, the therapy has been adapted so that it works well with people who have a language disability.

SUMMARY:
Around one third of stroke survivors will have aphasia, which means they will have difficulty talking, understanding, reading or writing. The main aims of this study are to assess: [1] the acceptability of an existing psychosocial intervention, solution focused brief therapy, to people with varying presentations of aphasia; and [2] the feasibility of conducting a future definitive trial investigating clinical and cost effectiveness.

DETAILED DESCRIPTION:
Background and Aims Around one third of people who have a stroke will experience aphasia, a language disability that can affect talking, understanding, reading or writing. The psychosocial impact of aphasia is considerable: those living with chronic aphasia are at risk of social isolation and depression. One potential intervention is Solution Focused Brief Therapy (SFBT). SFBT is an approach to building positive change in a person's life. It builds up a picture of a client's preferred future; encourages a person to notice positive signs of change; explores personal resources, skills and resilience; and acknowledges the impact of the stroke on a person's life and identity.

The current project builds on a small-scale proof-of-concept study that explored SFBT with five people who had mild to moderate aphasia, at least two years post stroke. There were improvements in participants' mood and participation and participants found the therapy highly acceptable.

The main aims of the current project are to assess: [1] the acceptability of SFBT to people with varying presentations of aphasia; and [2] the feasibility of conducting a future definitive trial investigating clinical and cost effectiveness.

Methods The overall study will last for 38 months (November 2016 to December 2019), and comprise a Development Phase (year 1) and a single-blind, randomized, wait-list controlled, feasibility trial with nested qualitative research comparing SFBT plus usual care to usual care alone (years 2 and 3).

During the Development Phase the investigators will develop the therapy manual and fidelity checking processes, train the clinicians, and finalize the protocol. Phase One has been informed through four workshops with the Aphasia Advisory Group, comprised of four people with aphasia and one carer, who advised on the study protocol and trial documentation. The investigators also conducted a pilot study with four people who have severe expressive and receptive aphasia where the investigators trialed the assessment and therapy protocol, and explored adapting the therapy for people with severe communication difficulties.

For the feasibility trial (commencing October 2017) 32 participants will be recruited with any severity of aphasia, at least six months post stroke. Participants will be randomly assigned to the intervention group or wait-list control group. Both groups will be assessed by a Research Assistant blinded to treatment allocation on psychosocial outcome measures at T1 (baseline, prior to randomization), T2 (three months post randomization) and T3 (six months post randomization). Participants will also take part in in-depth interviews at T3 exploring their experiences of taking part in the project as well as complete a resource use questionnaire. All participants will receive all usual care, and up to six SFBT sessions spaced over three months delivered by Speech and Language Therapists. The intervention group will receive the therapy immediately post randomization, while the wait-list control group will be offered the intervention after T3. The wait-list control will additionally be reassessed at T4 (nine months post randomization). The investigators will also interview the trial clinicians, and the Local Collaborators at the two participant identification sites.

Results The feasibility of recruitment and retention of participants (including proportion who consent; rate of consent; attrition rates) will be assessed, as will treatment fidelity. Descriptive statistics for the clinical outcome measures will be presented, for the entire trial population and by trial arm, at each time point, with means and confidence intervals plotted over time. The proportion of missing data will also be reported. As part of the economic evaluation, the relevant costs and health gains will be presented by trial arm and the completeness of data collection methods and their acceptability will be assessed. Qualitative data on acceptability of the intervention and study procedures will be analysed using Framework Analysis.

Clinical Implications This trial has been designed to assess the acceptability of the intervention for people with varying presentations of aphasia, and the feasibility of conducting a successful definitive trial evaluating clinical and cost effectiveness in the future. Given the high levels of distress and isolation experienced by people living with aphasia, and the current poor evidence base, there is a pressing need to investigate effective psychosocial interventions. SFBT is potentially a relatively brief approach deliverable by Speech and Language Therapists.

ELIGIBILITY:
Inclusion criteria:

* Have a diagnosis of ischaemic or haemorrhagic stroke
* At least six months post stroke
* 18 years old or over
* Presenting with aphasia as a result of the stroke. For those participants identified via United Kingdom National Health Service (two participant identification centers), this will be determined based on Speech and Language Therapist diagnosis. For participants recruited via the community, it will be based on their scores on the Frenchay Aphasia Screening Test (FAST). This test covers four major aspects of language: comprehension, expression, reading and writing. Aphasia is determined by published cut-off scores. Where a person has mild aphasia, such that they score as 'normal' on the FAST, but where the participant self-identifies as having aphasia, and this is confirmed by the clinical judgement of the Chief Investigator, they will be included.

Exclusion Criteria:

* Other diagnoses affecting cognition such as dementia or advanced Parkinson's Disease
* Severe uncorrected visual or hearing problems that would impact on a person's capacity to take part in the intervention
* Severe or potentially terminal co-morbidity on grounds of frailty
* Currently receiving a psychological or psychiatric intervention
* Non-fluent English speaker prior to the stroke based on self/family report
* Do not have mental capacity to consent to take part in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Warwick Edinburgh Mental Well-being Scale (WEMWBS) | 6 months post randomization
  Measures mental well-being. 14 items, scores range from 14 to 70, with higher scores indicating greater overall mental well-being

SECONDARY OUTCOMES:
Warwick Edinburgh Mental Well-being Scale (WEMWBS) - measuring change | All participants will complete WEMWBS at baseline, pre-randomization (T1), 3 months post randomization (T2), 6 months post randomization (T3). The wait-list control arm will also be tested at 9 months post randomization (T4).
  Measures mental well-being. 14 items, scores range from 14 to 70, with higher scores indicating greater overall mental well-being
General Health Questionnaire-12 (GHQ-12) - measuring change | All participants will complete GHQ-12 at baseline, pre-randomisation (T1), 3 months post randomisation (T2), 6 months post randomisation (T3). The wait-list control arm will also be tested at 9 months post randomisation (T4).
  Measures psychological distress. 12 items, scores range from 0 to 12 with higher scores indicating greater levels of distress
Communicative Participation Item Bank (CPIB) - measuring change | All participants will complete CPIB at baseline, pre-randomisation (T1), 3 months post randomisation (T2), 6 months post randomisation (T3). The wait-list control arm will also be tested at 9 months post randomisation (T4).
  Measures communicative participation. 10 items, scores range from 0 to 30 with higher scores indicating communication difficulties interfere less with participation
Depression Intensity Scale Circles (DISCS) - measuring change | All participants will complete DISCS at baseline, pre-randomisation (T1), 3 months post randomisation (T2), 6 months post randomisation (T3). The wait-list control arm will also be tested at 9 months post randomisation (T4).
  Measures depression. Single item scale, scores range from 0 to 5, with a score 0-1 indicating no/low distress, and 5 high distress; designed to be accessible to people with cognitive or communicative deficits.

OTHER OUTCOMES:
European Quality of Life - 5 dimensions, 5 levels (EQ-5D-5L) - measuring change | All participants will complete EQ-5D-5L at baseline, pre-randomisation (T1), 3 months post randomisation (T2), 6 months post randomisation (T3). The wait-list control arm will also be tested at 9 months post randomization (T4).
  Measures generic health status; the first part of the measure contains 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) that are rated on 5 levels (from no problems to extreme problems). The second part is a Visual Analogue Scale where a person self-rates their health. The EQ-5D-5L will be used to measure quality adjusted life years (QALYs) gained in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Northcott, PhD, Principal Investigator — City, University of London
Locations (1):
- City, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Northcott S, Thomas S, James K, Simpson A, Hirani S, Barnard R, Hilari K. Solution Focused Brief Therapy in Post-Stroke Aphasia (SOFIA): feasibility and acceptability results of a feasibility randomised wait-list controlled trial. BMJ Open. 2021 Aug 18;11(8):e050308. doi: 10.1136/bmjopen-2021-050308. PMID 34408055
- [Derived] Northcott S, Simpson A, Thomas S, Barnard R, Burns K, Hirani SP, Hilari K. "Now I Am Myself": Exploring How People With Poststroke Aphasia Experienced Solution-Focused Brief Therapy Within the SOFIA Trial. Qual Health Res. 2021 Sep;31(11):2041-2055. doi: 10.1177/10497323211020290. Epub 2021 Jun 15. PMID 34130554